CLINICAL TRIAL: NCT03291067
Title: A Randomized, Double Blind, Placebo Controlled Study to Assess the Effect of MT-8554 on the Frequency and Severity of Vasomotor Symptoms in Postmenopausal Women
Brief Title: MT-8554 for Reduction of Vasomotor Symptoms in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MT-8554-A01
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Results first posted 2022-01-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Menopause Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MT-8554 1mg (Experimental)
  Interventions: Drug: MT-8554 1mg
- MT-8554 5mg (Experimental)
  Interventions: Drug: MT-8554 5mg
- MT-8554 10mg (Experimental)
  Interventions: Drug: MT-8554 10mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-8554 1mg — MT-8554 1mg QD, oral, 12 weeks
  Arms: MT-8554 1mg
Drug: MT-8554 5mg — MT-8554 5mg QD, oral, 12 weeks
  Arms: MT-8554 5mg
Drug: MT-8554 10mg — MT-8554 10mg QD, oral, 12 weeks
  Arms: MT-8554 10mg
Drug: Placebo — Placebo QD, oral, 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of MT-8554 for treatment of vasomotor symptoms (VMS) associated with menopause.

DETAILED DESCRIPTION:
This is a Phase II randomized, double-blind, placebo-controlled study for dose selection in postmenopausal women with moderate to severe VMS, defined as follows:

* Moderate: sensation of heat with sweating, able to continue activity
* Severe: sensation of heat with sweating, causing cessation of activity This study is comprised of a screening period, a run-in period and a 12-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* Provide written informed consent to participate in this study
* Spontaneous amenorrhea for ≥12 months; or spontaneous amenorrhea for at least 6 months and with follicle stimulating hormone (FSH) levels >40 mIU/mL; or documented bilateral salpingo oophorectomy ≥6 weeks, with or without hysterectomy
* 7 or more moderate to severe VMS per day, or 50 or more moderate to severe VMS per week
* Have a consistent bedtime on at least 5 nights per week
* Mean VMS frequency during the Placebo Run in period does not drop by more than 50% from the mean level reported for 2 weeks during the Screening period
* VMS diary compliance >50%
* In the Investigator's opinion, subject is able to understand the nature of the study and any risk involved in participation, and is willing to cooperate and comply with the protocol restrictions and requirements

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* History of any cancer within 5 years except for basal cell carcinoma
* History of undiagnosed abnormal vaginal bleeding
* History of Hepatitis B, Hepatitis C or HIV
* History of psychiatric illness, excessive alcohol intake or use of recreational drugs who are unsuitable for study enrollment and compliance
* Presence or history of severe adverse reaction or allergy to any drug
* Peripheral vascular disease or disorders with associated vasculopathies
* Clinically significant conditions which could interfere with the objectives of the study or the safety of the subject, as judged by the Investigator
* Endometrial thickness of >=5 mm as measured by transvaginal ultrasound
* Abnormal result from baseline endometrial biopsy (i.e., endometrial hyperplasia or endometrial cancer)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin ≥2.0 × upper limit of normal (ULN) above the reference range
* Subjects of childbearing potential

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (53):
- United States (53):
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Norwalk, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, New London, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Wellington, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Sandy Springs, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Ankeny, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Marrero, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Morehead City, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Englewood, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Bristol, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Schertz, Texas
  - Research Site, Draper, Utah
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Covington, Washington
  - Research Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject with dual status of the run-in-failure and randomized in error in MT-8554 5 mg group was excluded from the Randomized Population.
Period: Overall Study
Arm/Group | MT-8554 1mg | MT-8554 5mg | MT-8554 10mg | Placebo
Started | 94 | 92 | 94 | 94
Treated | 95 | 90 | 93 | 90
Completed | 84 | 78 | 61 | 77
Not Completed | 10 | 14 | 33 | 17
Not completed — Adverse Event | 0 | 2 | 17 | 3
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 5 | 3 | 4 | 2
Not completed — Withdrawal by Subject | 3 | 4 | 7 | 5
Not completed — Other | 0 | 4 | 4 | 6

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants were number of participants who received at least one study medication which was indicated as "Treated" in the above Participant Flow module. 94 subjects were originally randomized to MT-8554 1mg group; but one subject in the placebo group took one week of MT-8554 1mg treatment in error. For calculation of "Treated" subjects, the subject was counted as MT-8554 1mg group so that "Treated" subjects in MT-8554 1 mg group was 95 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-8554 1mg | MT-8554 5mg | MT-8554 10mg | Placebo | Total
Number analyzed (Participants) | 95 | 90 | 93 | 90 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (6.27) | 54.6 (6.62) | 56.0 (6.55) | 55.7 (6.25) | 55.2 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 90 | 93 | 90 | 368
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 20 | 25 | 19 | 28 | 92
  White | 74 | 64 | 74 | 62 | 274
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Daily Frequency of Moderate to Severe VMS at Weeks 4 and 12
Description: The average daily frequency of moderate to severe VMS at a time point (Baseline, Weeks 4 and 12) was the average of the frequency of moderate to severe VMS of available diary days in a 7-day window. Changes in the average daily frequency of moderate to severe VMS at Week 4 and Week 12 compared to baseline were evaluated.
Time Frame: Baseline, Weeks 4 and 12
Population: Intent-to-treat (ITT) population=All randomized subjects who have at least 1 post-baseline efficacy assessment
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | MT-8554 1mg | MT-8554 5mg | MT-8554 10mg | Placebo
Number analyzed (Participants) | 93 | 90 | 89 | 91
VMS per day
  Week 4 | -1.92 (0.609) | -2.75 (0.705) | -2.75 (0.734) | -1.39 (0.705)
  Week 12 | -2.91 (0.690) | -3.11 (0.780) | -3.38 (0.821) | -2.78 (0.779)

2. Primary Outcome: Change From Baseline in the Average Daily Severity Score of Mild to Severe VMS at Weeks 4 and 12
Description: The daily severity score of VMS was defined as (2xFmo + 3xFse)/(Fmo + Fse) for baseline, and (1xFmi + 2xFmo + 3xFse)/(Fmi + Fmo + Fse) for Weeks 4 and 12, where Fmi, Fmo, and Fse were the daily frequencies of mild, moderate, and severe VMS, respectively. The average daily severity score of mild to severe VMS at a time point (Baseline, Week 4 and Week 12) was the average of the daily severity of available diary days in the corresponding 7-day window. The severity score of VMS ranged from 0 (lowest severity) to 3 (highest severity). Change in the average daily severity score of mild to severe VMS at Week 4 and Week 12 compared to baseline were evaluated.
Time Frame: Baseline, Weeks 4 and 12
Population: Intent-to-treat (ITT) population=All randomized subjects who have at least 1 post-baseline efficacy assessment
Measure: Least Squares Mean (Standard Error); unit: VMS severity score per day
Arm/Group | MT-8554 1mg | MT-8554 5mg | MT-8554 10mg | Placebo
Number analyzed (Participants) | 93 | 90 | 89 | 91
VMS severity score per day
  Week 4 | -0.302 (0.0609) | -0.407 (0.0714) | -0.305 (0.0740) | -0.316 (0.0712)
  Week 12 | -0.374 (0.0725) | -0.481 (0.0822) | -0.433 (0.0864) | -0.388 (0.0819)

3. Secondary Outcome: Percentage of Responders at Weeks 4 and 12
Description: Subjects with cutoff number or greater reduction in the average daily frequency of moderate and severe VMS compared to baseline. The cutoff number was calculated using anchor-based method. The cutoff number was defined as numerical value to maximize the sensitivity and the specificity, using Patient Global Impression of Change (PGIC) as the anchor.
Time Frame: Week 4 and Week 12
Population: Intent-to-treat (ITT) population=All randomized subjects who have at least 1 post-baseline efficacy assessment. The subjects without VMS frequency data at Week 4 were excluded from the analysis at Week 4. The subjects without VMS frequency data at Week 12 were excluded from the analysis at Week 12.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-8554 1mg | MT-8554 5mg | MT-8554 10mg | Placebo
Number analyzed (Participants) | 93 | 90 | 89 | 91
percentage of subjects
  Week 4: number analyzed (Participants) | 88 | 82 | 72 | 86
  Week 4 | 31.8 | 52.4 | 36.1 | 36.0
  Week 12: number analyzed (Participants) | 81 | 76 | 61 | 74
  Week 12 | 44.4 | 60.5 | 54.1 | 54.1

4. Secondary Outcome: Change From Baseline in the Insomnia Severity Index at Week 4 and Week 12
Description: The Insomnia Severity Index was a self-rated, 7-item validated sleep scale that measured clinical insomnia severity. The total score ranged from 0-28 where higher values indicated increased severity of insomnia.
Time Frame: Baseline, Weeks 4 and 12
Population: Intent-to-treat (ITT) population=All randomized subjects who have at least 1 post-baseline efficacy assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MT-8554 1mg | MT-8554 5mg | MT-8554 10mg | Placebo
Number analyzed (Participants) | 93 | 90 | 89 | 91
units on a scale
  Week 4 | -1.8 (0.49) | -3.1 (0.51) | -3.6 (0.55) | -1.8 (0.50)
  Week 12 | -3.2 (0.53) | -2.7 (0.55) | -2.4 (0.54) | -3.0 (0.55)

ADVERSE EVENTS:
Time Frame: Week 12
Description: One subject was randomized to placebo group; but the subject got one week of MT-8554 1 mg treatment so that the subject was counted as MT-8554 1 mg group in the Safety Population. Total of 6 subjects (3 on placebo, 2 on MT-8554 5 mg and 1 on MT-8554 10 mg) did not take any study medication so that these subjects were excluded from the Safety Population.
Arm/Group | MT-8554 1mg | MT-8554 5mg | MT-8554 10mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/90 | 0/93 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/95 | 1/90 | 0/93 | 0/90
Other Adverse Events (participants affected / at risk) | 37/95 | 41/90 | 46/93 | 37/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-8554 1mg (N=95) | MT-8554 5mg (N=90) | MT-8554 10mg (N=93) | Placebo (N=90)
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-8554 1mg (N=95) | MT-8554 5mg (N=90) | MT-8554 10mg (N=93) | Placebo (N=90)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 2 | 11 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 1
Cyst (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0
Feeling cold (General disorders) | 1 | 2 | 3 | 1
Feeling hot (General disorders) | 0 | 0 | 7 | 0
Feeling jittery (General disorders) | 0 | 1 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 2 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 3 | 1 | 2
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 1
Biopsy endometrium abnormal (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 4 | 1 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 1 | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 1 | 1 | 2
Blood urine present (Investigations) | 0 | 0 | 0 | 1
Body temperature decreased (Investigations) | 1 | 0 | 1 | 1
Electrocardiogram ST-T change (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 1
Low density lipoprotein increased (Investigations) | 2 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0
Oestradiol increased (Investigations) | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 1 | 1
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 3 | 1 | 1 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 5 | 0
Migraine (Nervous system disorders) | 2 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 14 | 2
Parosmia (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep inertia (Psychiatric disorders) | 0 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 2 | 0
Hot flush (Vascular disorders) | 1 | 0 | 3 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03291067/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03291067/SAP_001.pdf